CLINICAL TRIAL: NCT05051826
Title: Effect of 12-weeks Resistance Training in Water Combined With Land on Starting and Turning Performance of Chinese Adolescent Swimmer
Brief Title: Effect of Resistance Training in Water Combined With Land on Starting and Turning ,12-weeks Resistance Training
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universiti Putra Malaysia (Other)
Responsible Party: Principal Investigator, Guo Wei, Principal Investigator, Universiti Putra Malaysia
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Basic Science
Other Study IDs: Guo Wei
Record Dates: First submitted 2021-08-31; First posted 2021-09-21 (Actual); Last update posted 2021-09-21 (Actual); Status verified 2021-09

CONDITIONS: Resistance, APC
Keywords: Resistance training; Starting turning performance; Adolescent
MeSH Terms: conditions — Activated Protein C Resistance

STUDY DESIGN:
Intervention Model Description: In this experiment, the combination of water and land resistance training method was used to intervene the teenagers' turning and starting, and compared with the traditional strength training method
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 1.Drag Umbrella 2. Hand Resistance 3.Resistance Suit (Experimental): 1. In the water, a small umbrella is attached to the athlete to increase resistance.
  2. In the water, increase resistance by increasing the area of the hand.
  3. In the water, use swim shorts that increase resistance
  Interventions: Other: Resistance training that combines water and land
- 1 Resistance 2 Bands Swiss Ball 3 Medicine Ball 4 Pulley Pull (Experimental): 1. On land, use a stretch rope to increase resistance.
  2. On land, inflatable bouncy balls are used to increase strength.
  3. On land, solid balls are used to increase strength.
  4. On land, pulleys are used to increase resistance.
  Interventions: Other: Resistance training that combines water and land

INTERVENTIONS:
Other: Resistance training that combines water and land — Device: Swimmers in the experimental group received resistance training in water for 12 weeks, and the resistance training in the experimental group was divided into 3 categories:Resistance palm and resistance umbrella, resistance suit.
  Device: The swimmers in the experimental group underwent core strength training on land for 12 weeks, and the resistance training in the experimental group was divided into 4 types of resistance zones: Swiss ball, medicine ball and drive zone.The combination of two resistance training methods can improve teenagers' swimming performance.

SUMMARY:
Resistance training has been widely used in various sports and is a common practice aimed at improving competition performance, especially in swimming. Swimming performance is highly dependent on muscle strength, especially short distances. Water or land resistance training can improve the swimming performance, especially the swimming performance of 50 meters and 100 meters. Both type of training has their own strength and weakness. Hence, combining both methods strength may enhance swimmer performance. In addition, competitive swimming consists of different stages, namely start, clean swim, turn and finish. However, there is no literature on the influence of resistance training on starting and turning.

DETAILED DESCRIPTION:
Through experimental design and quantitative research methods. In this experiment, the resistance training method of water combined with land was used to intervene the turning and starting of young people, and the traditional strength training was compared to find out a better training method. The experiment will use 12 weeks of resistance training to improve the swimmer's turn and start intervention. The experiment consisted of four groups, 20 boys and 20 girls in the experimental group and 20 boys and 20 girls in the control group. Compare the differences between the two groups. Divided into discussion groups and general teaching groups. Two of the most significant differences, this experiment aims to provide a theoretical basis for improving the training methods of swimming, so that young swimmers can get better swimming performance, especially on the start and turn.

Experiment Group Week1-3: Drag Umbrella , Resistance Bands, Swiss Ball, Hand Resistance. Week3-6: Drag Umbrella , Resistance Bands, Swiss Ball, Hand Resistance. Week6-9: Drag Umbrella, Pulley Pull, Medicine Ball, Resistance Suit. Week9-12: Drag Umbrella Pulley Pull, Medicine Ball, Resistance Suit. Control Group Week1-3: Sit-Up, Press-Up, Deep Squat, Lift Heel Week 3-6: Sit-Up, Press-Up, Deep Squat, Lift Heel Week6-9: Dumbbell, Barbell ,Stomach Up, Squat Up Week9-12: Dumbbell, Barbell, Stomach Up, Squat Up

ELIGIBILITY:
Inclusion Criteria:

1. Swimmers participate in organized swimming training programs.
2. Participants with an average age of about 10 years.

Exclusion Criteria:

1. Untrained, novice, masters, and paraplegic swimmers.
2. Triathlon and water polo athletes.
3. Injured swimmers.

Ages: 10 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 80 (Actual)
Dates: Start 2021-02-09 (Actual); Primary Completion 2021-06-20 (Actual); Study Completion 2021-08-02 (Actual)

PRIMARY OUTCOMES:
starting and turning performance of Chinese adolescent swimmer | before the experiment
  Turning:
  1. Turn around time，（s）
  2. The time to swim to 5 meters, （s）
  3. The time to swim to 7 meters, （s）
  4. The time to swim to 10 meters，（s）
  Turning:
  1. Turn around time（s）
  2. The time to swim to 5 meters, （s）
  3. The time to swim to 7 meters, （s）
  4. The time to swim to 10 meters（s）
  Starting:
  1. The reaction time of the start（s）
  2. The time in the air, (Remove the backstroke)（s）
  3. The distance in the water, (Remove the backstroke)（m）
  4. The time to swim to 5 meters, （s）
  5. The time to swim to 7 meters, （s）
  6. The time to swim to 10 meters（s）

SECONDARY OUTCOMES:
starting and turning performance of Chinese adolescent swimmer | 6 weeks end
  Turning:
  1. Turn around time，（s）
  2. The time to swim to 5 meters, （s）
  3. The time to swim to 7 meters, （s）
  4. The time to swim to 10 meters，（s）
  Turning:
  1. Turn around time（s）
  2. The time to swim to 5 meters, （s）
  3. The time to swim to 7 meters, （s）
  4. The time to swim to 10 meters（s）
  Starting:
  1. The reaction time of the start（s）
  2. The time in the air, (Remove the backstroke)（s）
  3. The distance in the water, (Remove the backstroke)（m）
  4. The time to swim to 5 meters, （s）
  5. The time to swim to 7 meters, （s）
  6. The time to swim to 10 meters（s）

OTHER OUTCOMES:
starting and turning performance of Chinese adolescent swimmer | 12 weeks end
  Turning:
  1. Turn around time，（s）
  2. The time to swim to 5 meters, （s）
  3. The time to swim to 7 meters, （s）
  4. The time to swim to 10 meters，（s）
  Turning:
  1. Turn around time（s）
  2. The time to swim to 5 meters, （s）
  3. The time to swim to 7 meters, （s）
  4. The time to swim to 10 meters（s）
  Starting:
  1. The reaction time of the start（s）
  2. The time in the air, (Remove the backstroke)（s）
  3. The distance in the water, (Remove the backstroke)（m）
  4. The time to swim to 5 meters, （s）
  5. The time to swim to 7 meters, （s）
  6. The time to swim to 10 meters（s）

CONTACTS AND LOCATIONS:
Overall Officials: Wei Guo, Principal Investigator — University Putra Malaysia
Locations (1):
- Guo wei, Guyuan, Ningxia, China

IPD SHARING:
Plan to Share IPD: No
Since this is my doctoral thesis experiment, I won't share it until I graduate

REFERENCES:
- [Result] Crowley E, Harrison AJ, Lyons M. The Impact of Resistance Training on Swimming Performance: A Systematic Review. Sports Med. 2017 Nov;47(11):2285-2307. doi: 10.1007/s40279-017-0730-2. PMID 28497283
- See also: This article is from National Library of Medinice — http://pubmed.ncbi.nlm.nih.gov

DOCUMENTS (1):
  • Study Protocol (2021-08-10): https://cdn.clinicaltrials.gov/large-docs/26/NCT05051826/Prot_000.pdf